CLINICAL TRIAL: NCT06457503
Title: Single-Arm Study of Toripalimab in Combination With Cisplatin and Gemcitabine in Recurrent Metastatic Nasopharyngeal Carcinoma Systemic Treatment Naïve Participants
Brief Title: A Study of Toripalimab in Combination With Cisplatin and Gemcitabine in Participants With Recurrent Metastatic Nasopharyngeal Cancer
Acronym: TRANSPARENT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHS-007-01/RTOG 3521
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Nasopharyngeal Cancer Recurrent
Keywords: Programmed death 1 [PD1] inhibitor; Toripalimab; Recurrent metastatic nasopharyngeal cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — toripalimab; Cisplatin; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Toripalimab + cisplatin (or carboplatin) + gemcitabine (Experimental): Participants will receive the triple combination of cisplatin, gemcitabine and toripalimab (Chemotherapy-based treatment phase) followed by single-agent toripalimab (Maintenance treatment phase). The use of cisplatin can be substituted with carboplatin from cycle 2 onwards.
  Interventions: Drug: Toripalimab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Toripalimab — Participants will receive toripalimab via intravenous infusion (IV) on Day 1 every 3 weeks (Q3W) during the Chemotherapy-based treatment phase and Maintenance treatment phase.
  Other Names: JS001; TAB-001; CHS-007
Drug: Cisplatin — Participants will receive cisplatin via IV on Day 1 Q3W during the Chemotherapy-based treatment phase.
Drug: Gemcitabine — Participants will receive gemcitabine via IV on Day 1 and Day 8 Q3W during the Chemotherapy-based treatment phase.
Drug: Carboplatin — In the event of cisplatin-related nephrotoxicity or at the discretion of the investigator due to cisplatin-related poor tolerability, carboplatin can substitute for cisplatin use from cycle 2 onward. These participants will receive carboplatin via IV on Day 1 Q3W during the Chemotherapy-based treatment phase.

SUMMARY:
This study aims to investigate toripalimab with chemotherapy in participants with nasopharyngeal cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of toripalimab in combination with chemotherapy (cisplatin and gemcitabine), as measured by objective response rate (ORR) assessed by a Blinded Independent Central Review Committee (BICR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in first-line recurrent metastatic nasopharyngeal cancer participants (both Epstein-Barr virus (EBV) and non-EBV-associated).

ELIGIBILITY:
Key Inclusion Criteria:

* Histological or cytological confirmation of recurrent/metastatic nasopharyngeal cancer with either EBV or non-EBV-associated cancer. The following subgroups are included:

  * EBER/EBV-negative (HPV+/-)
  * EBER/EBV-positive (HPV+/-)
* Recurrent/metastatic (stage IV-B as defined by the International Union against Cancer [UICC] and American Joint Committee on Cancer [AJCC] staging system for nasopharyngeal cancer [NPC], eighth edition) or recurrent NPC after curative treatment. For recurrent NPC, more than 6 months between the last dose of radiotherapy or chemotherapy and the date of recurrence.
* Measurable disease based on RECIST v 1.1 as determined by the site. Note: Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

Key Exclusion Criteria:

* Disease that is suitable for local therapy administered with curative intent.
* Prior systemic therapy administered in the recurrent or metastatic setting. Participants who develop disease recurrence within 6 months from curative intent chemoradiation will be excluded.
* Rapidly progressing disease (e.g., tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
* Active or untreated central nervous system (CNS) metastases (e.g., brain or leptomeningeal), as determined on computerized tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments. Participants who have prior therapies for brain or leptomeningeal metastasis and have been stabilized ≥ 1 month and have discontinued systemic steroid therapy (>10 mg/day prednisone or equivalent) ≥ 1 month prior to enrollment are eligible.

Other protocol-defined inclusion and exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by a Blinded Independent Central Review (BICR) Committee according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 | Up to 24 months

SECONDARY OUTCOMES:
Duration of Response (DoR) assessed by BICR according to RECIST v1.1 | Up to 24 months
ORR assessed by the investigator according to RECIST v1.1 | Up to 24 months
DoR assessed by the investigator according to RECIST v1.1 | Up to 24 months
Progression-free Survival (PFS) assessed by BICR according to RECIST v1.1 | Up to 24 months
PFS assessed by the investigator according to RECIST v1.1 | Up to 24 months
Overall Survival (OS) defined as time from enrollment to death due to any cause | Up to 42 months
Disease Control Rate (DCR) assessed by BICR according to RECIST v1.1 | Up to 24 months
DCR assessed by the investigator according to RECIST v1.1 | Up to 24 months
Landmark PFS rates at 1 year and 2 years, derived from Kaplan-Meier (KM) curve | 12 months, 24 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - University of California, San Francisco, San Francisco, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Centre, Toronto, Canada